CLINICAL TRIAL: NCT06825390
Title: Mechanistic Clinical Trial of Auricular Stimulation and Cryogenic Auriculotherapy in Patients With Chronic Low-back Pain, Using Functional Near-infrared Spectroscopy and Magnetic Resonance Imaging
Brief Title: AuriculoTherapy NeuroImaging
Acronym: ATNI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keith M Vogt (Other)
Responsible Party: Sponsor-Investigator, Keith M Vogt, Associate Professor of Anesthesiology & Perioperative Medicine and Bioengineering, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY24090084
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain; Chronic Low-back Pain; Back Pain, Low; Lumbar Disc Disease; Lumbar Discogenic Pain; Lumbar Pain Syndrome; Lumbar Post-Laminectomy Syndrome; Back Pain Lower Back Chronic; Back Pain Without Radiation; Pain;Back Low;Chronic
Keywords: auriculotherapy; auricular stimulation; functional near-infrared spectroscopy; functional magnetic resonance imaging; functional connectivity; cryo-auriculotherapy
MeSH Terms: conditions — Low Back Pain; Intervertebral disc disease; Somatoform Disorders; post laminectomy syndrome; Back Pain

STUDY DESIGN:
Intervention Model Description: 1:1 randomized, double-blind, within-subject crossover design for mechanistic neuroimaging clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the investigator delivering the sham/verum auriculotherapy treatment will know the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active cryo-auriculotherapy first / sham second (Experimental): Participants randomly assigned to Group 1 will receive verum cryo-auriculotherapy treatment first, at the end of visit 1. They will return 5-7 days later for follow-up imaging (visit 2). After at least a 2 month wash-out period, all will return for their third visit, which will end with sham auricular intervention. Visit 4 is the second follow-up imaging session. All visits involve fNIRS imaging with auricular stimulation using von Frey filaments, prior to sham/cryo intervention.
  Interventions: Device: Cryo-auriculotherapy; Device: Sham auriculotherapy; Other: Experimental auricular stimulation
- Sham first / active cryo-auriculotherapy second (Experimental): Participants randomly assigned to Group 2 will receive sham auricular intervention first, at the end of visit 1. They will return 5-7 days later for follow-up imaging (visit 2). After at least a 2 month wash-out period, all will return for their third visit, which ends with verum cryo-auriculotherapy treatment. Visit 4 is the second follow-up imaging session. All visits involve fNIRS imaging with auricular stimulation using von Frey filaments, prior to sham/cryo intervention.
  Interventions: Device: Cryo-auriculotherapy; Device: Sham auriculotherapy; Other: Experimental auricular stimulation

INTERVENTIONS:
Device: Cryo-auriculotherapy — The cryo-IQ device (containing compressed nitrous oxide) with a narrow-tip nozzle will be used. After disinfection of the device and both ears, 7 inter-related points in the auricular cartography will be treated with a 1-2 second application of cold gas, applied to both ears. Treatment points will be: mesoderm master, spine, reticular formation, sensory master point, thalamus, adrenocorticotropic hormone, and corpus callosum.
Device: Sham auriculotherapy — For the sham procedure, an empty gas canister will be used in the cryo-IQ device. This will make the same noise and temporary skin imprint on the ear, but does not deliver any cooling effect. The same 7 ear points will be sham-treated in a protocol that is imperceptibly different from the verum auriculotherapy treatment.
Other: Experimental auricular stimulation — Three points on each ear will be repeatedly stimulated with a plastic (von Frey) filament. This will be felt, but not be painful and should not result in lasting irritation.
  Other Names: von Frey filament

SUMMARY:
This is a clinical study of patients who have low back pain (for at least 6 months). The goal is to understand, with brain imaging, how auriculotherapy (an acupuncture-like stimulation of the ear) may work to relieve pain. There are 4 total study visits, divided into two pairs of visits that occur before and 5-7 days after receiving either a real or sham auriculotherapy treatment. The cryo-IQ device will be used, to stimulate 7 small areas on both ears with a focused jet of cold as a small amount of compressed gas is released. This is generally not painful, and less invasive, compared to using needles for auriculotherapy.

DETAILED DESCRIPTION:
This is a 1:1 randomized, double-blind, sham-controlled, within-subject crossover trial of cyro-auriculotherapy in patients with chronic low back pain. Cryo-auriculotherapy is an effective alternative to needles, in which compressed gas provides focal (~1 mm2) persistent stim of auricular points, with minimal pain. Both before and 5-7 days after (time of peak effect) active vs. sham cryo-AT, resting brain connectivity will be measured with functional MRI and responses to a non-therapeutic experimental auricular stim paradigm (using von Frey filaments) will be recorded with functional near infra-red spectroscopy. After a 2-month washout period, patients will return for the same data collection surrounding the crossover intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, at least 18 years old
2. Episodes of chronic low back pain at least daily for at least 6 months, with an average pain score within the last week of 3/10.

Exclusion Criteria:

1. active lesions, skin disruptions, or neuropathy of either ear;
2. recent (<1 month) analgesic procedures or surgery;
3. recent (<1 month) start of new analgesic or psychoactive medication (including marijuana, opioids, tramadol, methadone, gabapentinoids, anti-depressants, anti-epileptics, mood-stabilizers, anti-psychotics, or stimulants);
4. history of chronic pain in shoulder or thumb (to avoid confounding at control stimulation points);
5. recent (< 3 months) illicit drug use;
6. prior substance misuse/abuse;
7. cold-activated diseases (including: agammaglobulinemia, cold urticaria, cold agglutinin disease, cryofibrinogenemia, cryoglobulinemia, immunosuppression, Raynaud's disease, collagen or autoimmune diseases, multiple myeloma, platelet deficiency disorders, pyoderma gangrenosum.)

   - MRI-specific exclusions additionally include:
8. Pregnancy or active attempts at conception;
9. Implanted metal or electronic device;
10. severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
functional near-infrared spectroscopy response, Lumbar spine vs. thumb auricular points | Baseline visit, over 10 minutes of data collection
  Calculated T-statistic for contrast of analyzed functional near-infrared spectroscopy (fNIRS) signal change, comparing responses from stimulation of the ipsilateral ear at the auricular points corresponding to the lumbar-spine vs. thumb. A T-statistic of 0 indicates no difference; more positive scores mean stronger fNIRS signal change with stimulation of the lumbar point, compared to stimulation of the thumb point; more negative scores mean change with stimulation of the thumb, compared to the lumbar spine. This outcome is a number reflecting the overall magnitude of difference between stimulation points, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.
Change in fNIRS response for Lumbar auricular point, for post- vs. pre- verum auriculotherapy, compared to post- vs. pre- sham auricular stimulation | Baseline, 5-7 days; 2 months, 9 weeks
  functional near-infrared spectroscopy data across the 4 sessions will be analyzed for double contrast: [(post-auriculotherapy treatment vs. pre-auriculotherapy treatment) minus (post-sham vs. pre-sham)], thus revealing significant differences in active treatment, compared to sham. The group-level T-statistic for the described contrast will be calculated from stimulation of the ipsilateral ear at the lumbar auricular point. The T-statistic is a single summary statistic reflecting the overall magnitude of differences in brain response to auricular stimulation after/before auriculotherapy treatment vs. sham. A T-statistic of 0 indicates no difference; larger positive values indicate a bigger difference in brain signal change after vs. before the active treatment, compared to after vs. before sham. Larger negative T-statistics indicate a larger change with sham, compared to active treatment. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.
Change in functional connectivity, for post- vs. pre- verum auriculotherapy, compared to post- vs. pre- sham auricular stimulation | Baseline, 5-7 days; 2 months, 9 weeks
  MRI data across the 4 sessions will be analyzed for changes in functional connectivity with the statistical comparison model: [(post-auriculotherapy treatment vs. pre-auriculotherapy treatment) minus (post-sham vs. pre-sham)], thus revealing significant differences in connectivity following the active treatment, compared to sham. A group-level T-statistic for the described contrast will be calculated from as a single summary statistic reflecting the overall magnitude of differences in brain connectivity change after/before auriculotherapy treatment vs. sham. A T-statistic of 0 indicates no difference; larger positive values indicate a bigger change in connectivity after vs. before the active treatment, compared to after vs. before sham. Larger negative T-statistics indicate a larger change with sham, compared to active treatment. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.

OTHER OUTCOMES:
Change in fNIRS response for Lumbar auricular point, for post- vs. pre- verum auriculotherapy, comparing male vs. female participants | Baseline, 5-7 days (before/after active treatment)
  fNIRS stimulation data from the after and before active auriculotherapy treatment will be analyzed for changes, performing a group level comparison between male and female participants. This will reveal sex-based differences in brain-response to auricular stimulation following auriculotherapy. A group-level T-statistic for the described contrast will be calculated from as a single summary statistic reflecting the overall magnitude of difference in brain response after/before auriculotherapy treatment for males vs. females. A T-statistic of 0 indicates no difference; larger positive values indicate greater change in response for males > females. Larger negative T-statistics will indicate a larger change in response for females > males. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.
Change in functional connectivity, for post- vs. pre- verum auriculotherapy, comparing male vs. female participants | Baseline, 5-7 days (before/after active treatment)
  MRI data from the after and before active auriculotherapy treatment will be analyzed for changes in functional connectivity, performing a group level comparison between male and female participants. This will reveal sex-based differences in response to auriculotherapy. A group-level T-statistic for the described contrast will be calculated from as a single summary statistic reflecting the overall magnitude of differences in brain connectivity change after/before auriculotherapy treatment for males vs. females. A T-statistic of 0 indicates no difference; larger positive values indicate greater change in connectivity for males > females. Larger negative T-statistics will indicate a larger change in connectivity for females > males. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Vogt, MD, PhD, Principal Investigator — University of Pittsburgh, UPMC
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be publicly shared, after deidentification.
Time Frame: De-identified individual participant data are anticipated to be available via open-access database within one year of study completion.
Access Criteria: This will be publicly available.